CLINICAL TRIAL: NCT02950363
Title: Assessment of Physician Mental Health Using Voice Analysis, Physiological Metrics and Smartphone Enabled Behavioral Modification
Brief Title: Physician Mental Health Study for Medical Trainees
Status: Completed | Type: Observational
Sponsor: Scripps Translational Science Institute (Other)
Collaborators: The Scripps Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-16-6803
Record Dates: First submitted 2016-07-06; First posted 2016-11-01 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-03

CONDITIONS: Mental Illness; Burnout Syndrome
Keywords: Depression; Suicide; Anxiety disorder; Burn out; Sleep quality; Stress
MeSH Terms: conditions — Mental Disorders; Burnout, Psychological; Depression; Suicide; Anxiety Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether use of a suite of smart phone enabled mobile health devices can reduce burnout in medical trainees. Such applications can then be used in more general populations with the same goal in mind.

DETAILED DESCRIPTION:
Wearable sensors and mental health platforms delivered via smartphones offer an opportunity to passively and actively acquire quantifiable signs and symptoms related to mental health status. These features include both physiological and cognitive performance measures. Collectively they serve as a set of metrics whereby an estimation of a person's mental state can be gauged. Additionally, use of these platforms allows those who are identified as high risk for mental illness to have targeted therapy delivered via their smartphone and if necessary connected with a suitable healthcare provider. Applications of such technology platforms serve to potentially reduce the substantial morbidity and mortality in a population at increased risk for mental illness and burnout.

ELIGIBILITY:
Inclusion Criteria:

* Trainee Physician at Scripps Green Hospital or Clinic.
* Older than 18 years.
* Must be reliable, cooperative and willing to comply with all protocol-specified procedures.
* Able to understand and grant informed consent
* Have a pre-existing smart phone capable of running all study software.

Exclusion Criteria:

* Has a significant medical condition that in the investigator's opinion may interfere with the study subject's optimal participation in the study.
* Known mental health condition including diagnosis of depression, schizophrenia, suicidality or anxiety disorder.
* Does not have suitable smart phone to allow all relevant software to run.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study is a single site prospective cross over observational study involving physicians at Scripps Clinic/Green Hospital, La Jolla, California. Subjects will serve as their own control group during a roll in phase of up to 3 months. All subjects will undergo at entry a baseline psychological survey (Maslach Burnout Index and PHQ-9). After the roll in phase, subjects will be provided with 3 smartphone-enabled devices (Oura Ring, Spire and Beyond Verbal voice analytics application). In addition to the devices, physicians will also be provided access to online educational content specific to physician burnout. Physicians will use the 3 devices for a 3 month period and Maslach Burnout Index and PHQ-9 assessments will be performed at a 6 week midpoint and at completion of the study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-07; Primary Completion 2017-05 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is change in Maslach Burnout Inventory (MBI) over a 16 week period as measured at time points Week 0 (Baseline), 4, 10, 16. | Week 0 (Baseline), 4, 10, 16
  Maslach Burnout Inventory

SECONDARY OUTCOMES:
Change in PHQ9 Score - (Raw score - No units) as measured at time points Week 0 (Baseline), 4, 10, 16. | Week 0 (Baseline), 4, 10, 16
  Change in PHQ9 Score over 3 months.
Relationship of absolute PHQ9 Score at weeks 4, 10 & 16 to a series of biometrics as described below: | Weeks 4, 10 & 16
  Average, following measurement of score:
  total time (Hours & Minutes) slept/night for week % sleep score (to Oura Ring App) per night for week min. overnight lowest heart rate (Beats per minute) per night for week
  Total time of per night for week:
  deep sleep (Hours & Minutes) light sleep (Hours & Minutes) REM sleep (Hours & Minutes) waking (Hours & Minutes) sleep latency (Hours & Minutes)
  % readiness score (% Measure native to Oura Ring App)
  Daily number of minutes of:
  focus (measured by Spire App) for week tension (measured by Spire App) for week calm (measured by Spire App) for week activity (measured by Spire App) for week inactivity (measured by Spire App) for week daily calories burned (measured by Spire App) for week
  Weekly # of (measured by the Beyond Verbal App):
  positive mood recordings negative mood recordings neutral mood recordings weekly arousal, temper, and valance score
Relationship of MBI score - 3 sub scales at weeks 4, 10 & 16 to a series of biometrics as described below: | Weeks 4, 10 & 16
  Average, following measurement of score:
  total time (Hours & Minutes) slept/night for week % sleep score (to Oura Ring App) per night for week min. overnight lowest heart rate (Beats per minute) per night for week
  Total time of per night for week:
  deep sleep (Hours & Minutes) light sleep (Hours & Minutes) REM sleep (Hours & Minutes) waking (Hours & Minutes) sleep latency (Hours & Minutes)
  % readiness score (% Measure native to Oura Ring App)
  Daily number of minutes of:
  focus (measured by Spire App) for week tension (measured by Spire App) for week calm (measured by Spire App) for week activity (measured by Spire App) for week inactivity (measured by Spire App) for week daily calories burned (measured by Spire App) for week
  Weekly # of (measured by the Beyond Verbal App):
  positive mood recordings negative mood recordings neutral mood recordings weekly arousal, temper, and valance score

CONTACTS AND LOCATIONS:
Locations (1):
- Scripps Health, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes